CLINICAL TRIAL: NCT02740465
Title: Anxiety and COPD Evaluation (ACE)
Brief Title: Anxiety and COPD Evaluation
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-00336
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: ACE; Anxiety; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD Patients (Experimental)
  Interventions: Behavioral: Anxiety Inventory for Respiratory Disease (AIR); Behavioral: Hospital Anxiety and Depression Scale (HADS)

INTERVENTIONS:
Behavioral: Anxiety Inventory for Respiratory Disease (AIR) — An initial version of the AIR was developed through a mixed-methods approach to item development, incorporating both emic and etic perspectives. This included an extensive review of extant anxiety scales (etic perspectives) and in-depth qualitative interviews with patients with COPD and self-reported anxiety (emic perspectives). AIR has ten items on a scale from 0 to 3. It provides a score of 0-30. High score indicates elevated level of clinically relevant anxiety symptoms.
Behavioral: Hospital Anxiety and Depression Scale (HADS) — The Hospital Anxiety and Depression Scale (HADS), a self-assessment scale, was developed to detect states of depression, anxiety and emotional distress amongst patients who were being treated for a variety of clinical problems.

SUMMARY:
This prospective, multicenter, cohort study is designed to validate Anxiety Inventory Respiratory Disease questionnaire in patients with Chronic Obstructive Pulmonary Disease (COPD).

The primary purpose of this study is to assess the validity of the Anxiety Inventory Respiratory (AIR) scale in detecting anxiety in relation to the DSM-V criteria in patients with COPD.

* To evaluate associations between COPD symptom scores assessed by the CAT questionnaire and MMRC dyspnea scale and measures of depression and anxiety
* To evaluate associations between physiologic measures of lung function (spirometry) and exercise tolerance (6 minute walk) and measures of depression and anxiety
* To evaluate associations between exacerbations of COPD and the prevalence of anxiety and depression in a cohort of COPD patients

DETAILED DESCRIPTION:
The goal of the Anxiety and COPD Evaluation (ACE) study is to validate the AIR scale by employing the Mini International Neuropsychiatric Interview to identify anxiety in 200 patients recruited at participating centers from the American Lung Association (ALA) Airways Research Network.

Confidential, not

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilation FEV1 < 80% of the predictive normal value and FEV1 (forced expiratory volume in one second) / Forced vital capacity(FVC) ratio < 0.7
* Clinically stable COPD as defined by stable maintenance of COPD medications and absence of an exacerbation of symptoms requiring treatment with an antibiotic or corticosteroids

Exclusion Criteria:

* Exacerbation of respiratory symptoms in the past six weeks that resulted in the need for treatment or hospitalization
* Unstable coronary heart disease such as recent myocardial infarction (within 3 months), untreated arrhythmia, or unstable angina
* Major psychiatric disorders (except for depression and anxiety disorders) such as schizophrenia, schizoaffective, or other disorders that in the opinion of the study physician that would affect study participation
* Montreal Cognitive Assessment (MoCA) < 18
* Disease or condition expected to cause death within six months or inability to perform study procedures, as judged by study physician

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 10 Minutes
  The Montreal Cognitive Assessment (MoCA) was developed as a brief screening instrument to detect mild cognitive impairment. It is a paper-and-pencil tool that requires approximately 10 minutes to administer, and is scored out of 30 points. The MoCA assesses multiple cognitive domains including attention, concentration, executive functions, memory, language, visuospatial skills, abstraction, calculation and orientation. It is widely used around the world and is translated to 36 languages and dialects.
COPD Assessment Test (CAT) | 10 Minutes
  The CAT is an eight-item questionnaire designed to quantify the impact of COPD symptoms on the health status of patients. The CAT is quick and easy for patients to complete and, without complex calculations, provides a score of 0-40 to indicate the impact of disease.
Modified Medical Research Council dyspnea scale (MMRC) | 10 Minutes
  The MMRC uses a simple grading system to assess a patient's level of dyspnea and has been used for many years for grading the effects of breathlessness on daily activities. This scale has been particularly used in patients with chronic obstructive pulmonary disease (COPD) in whom it has proved to be useful and complementary to First Forced expiratory volume (FEV1) in the classification of disease severity.
Pittsburgh Sleep Quality Index (PSQI) | 1-month time interval
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Patient-Reported Outcomes Measurement Information System Questionnaires: Emotional Distress-Anxiety Function -(PROMIS-29) | 10 Minutes
  These patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. The NIH funded leading PRO and clinical investigators to develop a "psychometrically validated, dynamic system to measure PROs efficiently in study participants with a wide range of chronic diseases and demographic characteristics." The PROMIS initiative is part of the NIH goal to develop systems to support NIH-funded research supported by all of its institutes and centers. PROMIS measures cover physical, mental, and social health and can be used across chronic conditions.
Patient-Reported Outcomes Measurement Information System Questionnaires: Physical Function - Short Form 20a (PROMIS-20a) | 10 Minutes
EuroQol EQ-5D- 5L | 10 Minutes
  The EQ-5D-5L is a generic measure of health related quality of life that can be calibrated on a 0 to 1 scale and thus measures utility, allowing for the calculation of Quality Adjusted Life Years (QALYs). The standard EQ-5D measures 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression graded from level 1 (i.e., no problems) to level 5 (i.e., extreme problems). Use of the 5-levels (EQ-5D-5L) rather than the standard 3 level EQ-5D (EQ-5D-3L) has led to less ceiling effect, greater discriminative ability, and potentially more power to detect differences between groups compared with EQ-5D-3L.
Patient Health Questionnaire for Depression (PHQ9) | 2 Days
  The Patient Health Questionnaire is a diagnostic tool for mental health disorders used by health care professionals that is quick and easy for patients to complete.
Patient Health Questionnaire for Anxiety (GAD7) | 2 Days
  A brief scale for anxiety and scores seven common anxiety symptoms.
Hospital Anxiety and Depression Scale (HADS) | 2 Days
  The Hospital Anxiety and Depression Scale (HADS), a self-assessment scale, was developed to detect states of depression, anxiety and emotional distress amongst patients who were being treated for a variety of clinical problems.
Mini International Neuropsychiatric Interview (MINI) | 10 Minutes
  Participants will be interviewed for unipolar major depression and anxiety disorders using the MINI, version 7.0 which conforms to the Diagnostic and Statistical Manual of Mental (DSM) Disorders.
6 Minute Walk Distance | 6 Minutes
  The purpose of the six minute walk is test exercise tolerance in chronic respiratory disease and heart failure. The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in that time. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Pulmonary function Spirometry pre and post bronchodilator | 2 Days
  Spirometry is a common office test used to diagnose asthma, chronic obstructive pulmonary disease (COPD), and certain other conditions that affect breathing. Spirometry measures how much air inhaled and exhaled and how fast.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Reibman, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States